CLINICAL TRIAL: NCT05722639
Title: Evaluation of Accuracy and Consistency of the X-Trodes System
Status: Completed | Type: Observational
Sponsor: B-Cube (Other)
Collaborators: X-Trodes (Unknown)
Responsible Party: Principal Investigator, Moran Cerf, Professor, B-Cube
Other Study IDs: Pro00068380
Record Dates: First submitted 2023-01-23; First posted 2023-02-10 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Equipment and Supplies
Keywords: Electrophysiology; Electrooculography; Electromyography; Electrocardiogram; Device; Acquisition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Representative sample of the U.S. population: Subjects will be fitted with two electrophysiology acquisition systems (one is FDA-approved, and the other is the one evaluated).
  Signals from both systems will be acquired simultaneously while the subjects rest and perform no cognitive tasks.
  Following, the signals from both devices will be assessed by an electrophysiology expert to determine if they are of equal quality.
  Interventions: Device: X-Trodes acquisition system

INTERVENTIONS:
Device: X-Trodes acquisition system — No intervention. The participants will sit passively while electrophysiology signals are captured from two devices in order to evaluate the signal quality.

SUMMARY:
The purpose of this study is to evaluate the accuracy and consistency of the X-Trodes acquisition system compared to a Food and Drug Administration (FDA)-cleared clinical electrophysiology device.

DETAILED DESCRIPTION:
The study aims to demonstrate that the performance of the study X-Trodes acquisition system is equivalent to that of an FDA-cleared clinical electrophysiology devices (in measuring electroencephalography , electrooculography, electromyography, and electrocardiogram signals).

Subjects will wear both devices simultaneously while signals are captured in resting state. Following, an evaluation of the similarity of signals between the two devices will be conducted. The evaluation will determine if the quality of the X-Trodes system matches that of the FDA-approved device.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, subjects must meet all the following inclusion criteria:

* Adults (age 21 - 99)
* Referred to an electrophysiology test by either neurologist or cardiologist in the last 5 years
* Produce interpretable electrophysiological signals by the acquisition devices

Exclusion Criteria:

* Did not sign the informed consent
* Cannot maintain the electrodes attached to their skin (i.e., due to beard on the chin area)
* Diagnosed as suffering from sleep apnea
* Pregnant or lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals ages 21 and over who are able to come to the study site and sit for about 30 minutes while two electrophysiology devices are capturing EEG, EOG, EMG, ECG signals from their body. Subjects should have no beard (to ease the signal capturing), not be pregnant, not suffer from sleep apnea, and comfortable with the study protocol (i.e., sign a consent form).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Signals alignment between two devices | Within 3 months from the completion of data collection.
  Electrophysiological time-series (EEG, EOG, ECG, EMG) in 2 recorded devices will be compared.
  For each subject, the time-series from 2 devices will be assessed by three independent raters (US board-certified neurologist/cardiologist). The raters will rank the quality of signals (1-signal is corrupt or unusable; 5-signal is clean and useable). Raters will be blind to the signal device.
  Time-series will be deemed interpretable if at least 2 of the raters scored it 4-5.
  Following the rater evaluation, the outcome will also be reported as a binary output where scores of 4-5 are considered interpretable signals.
  The trial will be considered successful if the number of high-quality (mean score 4-5) X-Trode series will be within one-standard deviation from the FDA-approved device's series while both systems yield over 80% high-quality signals.
Assessment of agreement among raters | Within 3 months from the completion of data collection.
  Agreement among raters will be evaluated by calculating the Intraclass correlation coefficient (ICC). ICC will be calculated for each of the 4 electrophysiological modalities. The acceptance criterion for ICC is 0.60 and higher.
  If no agreement among rates is observed (ICC < 0.6) then Spearman correlation coefficient between each pair of raters for the specific signal (per subect, per time-series) will be calculated and the rankings of the two raters with the highest correlation coefficient will be selected for the analysis.

OTHER OUTCOMES:
Subjects descriptive statistics | 1 month after completion of data collection.
  Description of subjects demographics, age, race, and gender will be reported.
Signal descriptive statistics | 1 month after completion of data collection.
  For the continuous electrophysiological data collected, summary table with sample size, mean, standard deviation of the signal for each subject and for the entire subjects cohort, median activity for each individual signal electrophysiological time-series, minimum, and maximum values will be reported.
Study descriptive statistics | 1 month after completion of data collection.
  ounts and percentage of any adverse events by type (ADE, SADE, ASADE, and USADE/UADE) will be tabulated.

CONTACTS AND LOCATIONS:
Locations (1):
- B-Cube, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No